CLINICAL TRIAL: NCT00427037
Title: Efficacy of Cholecalciferol (Vitamin D3) Therapy in Correcting Vitamin D Insufficiency and Secondary Hyperparathyroidism in Subjects With Chronic Kidney Disease: A Randomized, Placebo Controlled Pilot Study
Brief Title: Cholecalciferol (Vitamin D3) Therapy in Chronic Kidney Disease (CKD) Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlanta VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Vin Tangpricha, Principal Investigator, Atlanta VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vitamin D-2006
Record Dates: First submitted 2007-01-24; First posted 2007-01-26 (Estimated); Results first posted 2009-03-12 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Kidney Disease; Vitamin D Deficiency
Keywords: Vitamin D deficiency; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Cholecalciferol (Active Comparator): D3
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — 50,000 IU weekly by mouth
  Other Names: Vitamin D3 is cholecalciferol
  Arms: Cholecalciferol
Drug: Placebo — identical placebo pill orally by mouth
  Other Names: D3
  Arms: Placebo

SUMMARY:
This is a 12 week pilot and feasibility study with an enrollment goal of 30 subjects. Half of the subjects will be randomized to vitamin D3 and the other half will receive a placebo. Subjects will be referred from the nutrition or renal clinic at Emory. CKD stage 3 and 4 patients will be eligible for participation if they have been determined to have vitamin D deficiency and are not on treatment with vitamin D or vitamin D analogues. Subjects will sign an informed consent form after reviewing the protocol in detail with the principal investigator. A questionnaire would collect information about dietary vitamin D intake, sunlight exposure, and any symptoms of vitamin D deficiency. The subject will have baseline levels of serum vitamin D (25-hydroxyvitamin D), parathyroid hormone (PTH), serum calcium and phosphate, creatinine and other markers of bone turnover. The questionnaires and the blood draws would be repeated on the 6th and 12th week of the study. Subjects will be given 12 pills of each containing either 50,000 IU vitamin D or placebo and asked to take one pill a week. They would be scheduled to return to the clinic after 6 weeks and blood measurements would be repeated. Subjects will be asked to revisit for their final visit at the 12th week when they would have their last blood draw and assessment.

DETAILED DESCRIPTION:
Vitamin D supplementation in reducing secondary hyperparathyroidism in chronic kidney disease patients, stage 3 and 4: A randomized, placebo controlled pilot study Problem of interest Chronic Kidney Disease (CKD) patients suffer from severe metabolic bone disease, which represents a formidable challenge to physicians. Defective vitamin D metabolism, and secondary parathyroid activation have been suggested as possible causes. Vitamin D is important for musculoskeletal health. Vitamin D can be obtained from the diet or made in the skin from exposure to sunlight, but it has to be converted by the kidneys into calcitriol, the active form in order to be effective. Decreased kidney mass in CKD patients causes reduced capability to convert vitamin D into calcitriol due to less 1-alpha hydroxylase enzyme levels. Current standard of care for patients with chronic renal disease is treatment with vitamin D analogues such as Rocaltrol or Hectoral. However, these medications have the potential to cause hypercalcemia. Studies have shown that calcitriol production becoming dependent on 25- hydroxyvitamin D availability in moderate CKD patients. There is speculation that there is still some "reserve" left for the generation of calcitriol from vitamin D in these patients.

The main question being posed in this study is:

Primary: Can a weekly high dose supplementation of cholecalciferol be effective in raising 25(OH)D levels in patients with CKD and can this reduce parathyroid hormone levels in pre-dialysis chronic kidney disease patients?

Study Design This is an 12 week pilot and feasibility study with an enrollment goal of 30 subjects. Half of the subjects will be randomized to vitamin D3 and the other half will receive a placebo. Subjects will be referred from the nutrition or renal clinic at Emory. CKD stage 3 and 4 patients will be eligible for participation if they have been determined to have vitamin D deficiency and are not on treatment with vitamin D or vitamin D analogues. Subjects will sign an informed consent form after reviewing the protocol in detail with the principal investigator. A questionnaire would collect information about dietary vitamin D intake, sunlight exposure, and any symptoms of vitamin D deficiency. The subject will have baseline levels of serum vitamin D (25-hydroxyvitamin D), parathyroid hormone (PTH), serum calcium and phosphate, creatinine and other markers of bone turnover. The questionnaires and the blood draws would be repeated on the 6th and 12th week of the study. Subjects will be given 12 pills of each containing either 50,000 IU vitamin D3 or placebo and asked to take one pill a week. They would be scheduled to return to the clinic after 6 weeks and blood measurements would be repeated. Subjects will be asked to revisit for their final visit at the 12th week when they would have their last blood draw and assessment.

Treatment This is a randomized control trial. Only half of the subjects will receive vitamin D treatment and the other half placebo. If at the end of the study, the subject is still vitamin D deficiency, they will be referred to an endocrinologist or to their primary doctor for treatment.

Scientific advancement If successful, this study would provide the necessary preliminary data in order to conduct a larger randomized controlled study supplementing vitamin D in chronic kidney disease patients. One potential area of study would be to see whether subjects supplemented with vitamin D were able to raise their active vitamin D levels using the "reserve" hydroxylase enzyme in the kidneys compared to those subjects who were just supplemented with a placebo. This study is necessary in order to determine whether weekly intake of a high dose vitamin D is sufficient to decrease the parathyroid hormone levels in the given time frame.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85
* CKD stage 3-4 (GFR 15-59 ml/min/1.73 m2 body surface area, calculated by using the MDRD Study equation GFR Calculator)
* serum 25(OH)D concentrations ≤ 30 ng/mL, and serum PTH levels >70 pg/mL documented within the last six months

Exclusion Criteria:

* History of liver failure (serum AST or ALT > 3-fold the upper limit of normal)
* requiring dialysis at any stage of the study
* history of intestinal malabsorption or chronic diarrhea
* serum calcium level (corrected for serum albumin) > 10.5 mg/dL
* calcium x phosphorus product >70
* treatment with more than 1000 IU of vitamin D per day, or current treatment with a vitamin D analogue or calcimimetic
* an anti-epileptic medication and other medications which can affect vitamin D metabolism (e.g., phenobarbital, phenytoin, rifampicin)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-12; Primary Completion 2006-07 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vin Tangpricha, M.D. Ph.D., Principal Investigator — Emory University
Locations (1):
- Emory Clinic, Atlanta, Georgia, United States

REFERENCES:
- [Result] Chandra P, Binongo JN, Ziegler TR, Schlanger LE, Wang W, Someren JT, Tangpricha V. Cholecalciferol (vitamin D3) therapy and vitamin D insufficiency in patients with chronic kidney disease: a randomized controlled pilot study. Endocr Pract. 2008 Jan-Feb;14(1):10-7. doi: 10.4158/EP.14.1.10. PMID 18238736
- [Derived] Alvarez JA, Law J, Coakley KE, Zughaier SM, Hao L, Shahid Salles K, Wasse H, Gutierrez OM, Ziegler TR, Tangpricha V. High-dose cholecalciferol reduces parathyroid hormone in patients with early chronic kidney disease: a pilot, randomized, double-blind, placebo-controlled trial. Am J Clin Nutr. 2012 Sep;96(3):672-9. doi: 10.3945/ajcn.112.040642. Epub 2012 Aug 1. PMID 22854402
- See also: Medscape Link — http://www.medscape.com/viewarticle/572253_1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study subjects were recruited from Nephrology and Endocrinology clinics at Emory University School of Medicine
Groups:
- Placebo: This is a matching placebo
- Cholecalciferol: This is vitamin D3 or Cholecalciferol
Period: Overall Study
Arm/Group | Placebo | Cholecalciferol
Started | 17 | 17
Completed | 10 | 10
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cholecalciferol | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (10.4) | 62.2 (11) | 60.8 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Secondary Outcome: Bone Turnover Marker-CTX
Description: Blood levels of C-telopeptide
Time Frame: 12 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Placebo | Cholecalciferol
Number analyzed (Participants) | 8 | 9
pg/mL | 0.24 [0.14 to 0.4] | 0.29 [0.18 to 0.49]

2. Primary Outcome: 25-hydroxyvitamin D
Description: 25-hydroxyvitamin D measured in serum by ELISA
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Placebo | Cholecalciferol
Number analyzed (Participants) | 10 | 10
ng/mL
  Baseline | 18.6 [12.8 to 27.1] | 17.3 [11.8 to 25.2]
  12 weeks | 19.5 [13.4 to 28.4] | 49.4 [33.9 to 72]

ADVERSE EVENTS:
Time Frame: 3 Months
Arm/Group | Placebo | Cholecalciferol
Serious Adverse Events (participants affected / at risk) | 1/17 | 1/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | Cholecalciferol (N=17)
Death (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes